CLINICAL TRIAL: NCT05827744
Title: The Evaluation of the Relationship Between Thicknesses and Isokinetic Strength of Hip Flexor and Extensor Muscles in Patients With Unilateral Traumatic Transfemoral Amputation
Brief Title: The Relationship Between Thicknesses and Isokinetic Strength of Hip Flexor and Extensor Muscles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 36
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Amputation, Traumatic
Keywords: amputation; hip flexors; hip extensors
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Isokinetic evaluations — Peak torque and total amount of work of hip flexors and extensors will be determined by the Cybex 6000 model computer-aided isokinetic system.
Other: Ultrasonographic evaluations — Ultrasonographic evaluations will be performed with a 5-12 MHz linear probe (Logic e portable; GE Healthcare, China). The thicknesses of the hip flexor (psoas major) and extensor (gluteus maximus) muscles will be measured while the patient is in the prone position, in accordance with the literature.

SUMMARY:
The aim of this study is to investigate the relationship of hip muscle thicknesses measured by ultrasonography with hip flexion and extension strength and clinical parameters in prosthesis users with unilateral traumatic transfemoral amputation.

DETAILED DESCRIPTION:
The aim of this study is to investigate the relationship of hip muscle thicknesses measured by ultrasonography with hip flexion and extension strength and clinical parameters in prosthesis users with unilateral traumatic transfemoral amputation.

This study will be useful in understanding whether ultrasonography is an appropriate imaging method in the follow-up of changes in functional strength in the hip girdle in patients with unilateral traumatic transfemoral amputation.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65
* The time elapsed after amputation > 6 months
* Using prosthesis for at least 3 months
* Being able to walk without an assistive device

Exclusion Criteria:

* Bilateral lower extremity amputation
* Presence of neurological, cardiovascular, and pulmonary disease that may affect walking performance

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 27 patients with unilateral transfemoral amputation
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
6-minute walking test (6MWT) | through study completion, an average of one month
  Functional performance will be assessed by 6MWT (in meter). Patients will be instructed to walk quickly, safely, and as much distance as possible over a rectangular path.
10-meter walking test | through study completion, an average of one month
  The short-distance over-ground gait speed will be assessed using a 10-Meter Walk Test. Participants will be asked to walk at normal pace on a 10-meter walkway.
Timed up and go test | through study completion, an average of one month
  Timed up and go test will be used for quantifying functional mobility balance. Participants will be instructed to sit in a comfortable position on a 45-65 cm high steady chair with a backrest and armrest, with both arms resting on their thighs, and then quickly stand up and move towards and around a fixed cone 3 m away, return, and sit again.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Örücü Atar, Principal Investigator — assistant professor
Locations (1):
- Ankara Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)